CLINICAL TRIAL: NCT01352819
Title: A Post Market Clinical Evaluation of Deep Brain Stimulation as an Adjunctive Treatment for Reducing Some of the Symptoms of Advanced, Levodopa-responsive Parkinson's Disease That Are Not Adequately Controlled With Medication
Brief Title: Post Market (Libra/LibraXP System) Deep Brain Stimulation (DBS) Parkinson's Disease Study
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: NM-09-036-EU-DB
Record Dates: First submitted 2011-04-14; First posted 2011-05-12 (Estimated); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The objective of this study is to evaluate the effectiveness of Deep Brain Stimulation as an adjunctive treatment for reducing some of the symptoms of advanced, levodopa-responsive Parkinson's disease that are not adequately controlled with medication.

It is the first study in Parkinson patients outside the US with a Deep Brain Stimulation system using constant current instead of constant voltage and using a lead with an active electrode tip.

DETAILED DESCRIPTION:
This study is designed as a prospective, observational, non-randomized, multi-centered study for 12 months in duration from implantation with the subjects being used as their own control. The primary outcome assessment will occur at three months: however, subjects will be followed for one year.

A comparison of measures within the same person from pre-treatment to post-treatment will be performed. Also, pre-treatment and post-treatment group means and standard deviations will be determined.

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in this study must meet the following inclusion criteria:

1. Subject has signed an informed consent.
2. Subject has been diagnosed, by a neurologist, with idiopathic Parkinson's disease.
3. Subject is a candidate for surgery.
4. Subject is 18 to 80 years of age.
5. Subject has a history of improvement of Parkinson's symptoms as a direct result of administering l-dopa to the subject with at least a 25% improvement in Unified Parkinson's Disease Rating Scale (UPDRS) motor score or subject has been diagnosed with tremor-dominant Parkinson's disease.
6. Subject should be stable on anti-Parkinson's disease medication for at least one month prior to study enrollment.

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the following criteria:

1. Subject has any major illness or medical condition that in the opinion of the physician would interfere with participation in the study.
2. Subject has non-treated clinically significant depression or any other significant psychiatric co-morbidities.
3. Subject has any condition requiring repeated MRI scans;
4. Subject has any condition requiring diathermy;
5. Subject is on anticoagulant medications and is unable to interrupt for time of procedure.
6. Subject has a history of cranial surgery.
7. Subject has dementia that interferes with their ability to co-operate or comply with study requirements or comprehend the Informed Consent as determined by the investigator.
8. Subject abuses drugs or alcohol.
9. Subject has a history of seizure
10. Subject has confirmation of diagnosis of a terminal illness associated with survival <12 months.
11. Female that is lactating or of childbearing potential with positive urine pregnancy test or not using adequate birth control.
12. Subject has participated in a drug, device or biological trial within the preceding 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Libra™/LibraXP™ DBS System Eligible subjects in this study will be screened to confirm that they meet the strict guidelines for advanced, levodopa-responsive Parkinson's disease that are not adequately controlled with medication followed by surgery to implant the Libra™/LibraXP™ deep brain simulation system.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2011-05; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
UPDRS motor scores | [Time Frame: 3 months after device implantation].
  Comparison of Parkinson's symptoms as demonstrated by the UPDRS motor scores in the medication 'Off' state at Baseline compared to the medication 'Off' with stimulation "On" 3 months after device implantation

SECONDARY OUTCOMES:
Satisfaction of therapy | [through 3, 6 months and 1 year]
  Rate of subject and caregivers therapy satisfaction through 3, 6 month and 1 year
Economic burden of the disease | [at baseline and 1 year]
  Rate on economic burden of the disease for caregiver determined from economic burden questionnaire at baseline and 1 year
Rating on caregiver's burden determined from Zarit Caregivers Burden Interview (ZCBI) | [at baseline, 3 month and 1 year]
Assessment of the way of coping as determined from the Way of Coping Checklist (WCC) from caregiver | [baseline, 3,6 month and 1 year]

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vesper, Prof, Principal Investigator — Universitätsklinukum Dusseldorf
Locations (6):
- France (2):
  - Hopital Neurologique, Lyon
  - CHU Laennec, Nantes
- Germany (3):
  - University Hospital Bonn, Bonn
  - University Hospital of Duesseldorf, Düsseldorf
  - University Hospital Regensburg, Regensburg
- Erciyes University Medicine School, Kayseri, Turkey (Türkiye)